CLINICAL TRIAL: NCT01499901
Title: Interest of the Bilateral Cochlear Implantation in the Deep Deaf Children Respect to the Unilateral Implantation - a Randomized Test
Brief Title: Comparison of the Bilateral Sequential and Simultaneous Cochlear Implantation in the Deaf Children
Acronym: Cochleo
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Recommendations of HAS have changed, the study is now useless
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P091204; HAO 09048 (Other: Assistance Publique)
Record Dates: First submitted 2011-12-06; First posted 2011-12-26 (Estimated); Last update posted 2012-11-19 (Estimated); Status verified 2012-11

CONDITIONS: Deafness
Keywords: deafness; unilateral implantation; bilateral; auditory perception
MeSH Terms: conditions — Deafness

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- sequential (Experimental): implantation bilateral sequential
  Interventions: Procedure: bilateral cochlear Implantation in sequential
- simultaneous (Experimental): implantation bilateral simultaneous
  Interventions: Procedure: bilateral cochlear Implantation in simultaneous

INTERVENTIONS:
Procedure: bilateral cochlear Implantation in sequential — bilateral cochlear Implantation in sequential
  Arms: sequential
Procedure: bilateral cochlear Implantation in simultaneous — bilateral cochlear Implantation in simultaneous
  Arms: simultaneous

SUMMARY:
In France the indication of bilateral cochlear implant (CI) is limited to specific cases. The impact on perception and language of bilateral CI simultaneous versus sequential has to be established before discussing the enlargement of indications.

DETAILED DESCRIPTION:
French multicentric study. 100 children, profound, congenitally deaf, aged between 10 months and 40 months, with indication of unilateral CI will be included. Randomization: 50 sequential at one year CI versus 50 simultaneous bilateral CI, their results compared. Main measures at 12 and 24 months: speech perception in silence and in noise. Other measures: sound localisation, oral language, vestibular impact, quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Deep bilateral congenital deafness.
* Age at the implantation: from 10 to 40 months, included.
* Criteria for indication of unilateral implantation (those considered by the HAS (2007))
* Deep bilateral deafness
* Threshold prosthetic equal or above 60 dB
* Intelligibility test in open list, below 30%, (to children under 3 years old : raw score in the questionnaire of the M.A.I.S. (72) below 15 with 2 apparatus)
* No medical nor radiologic contraindication
* Entitled child for welfare (excepted medical state aids)
* French spoken at home
* Agreement firms for the study by the two genitors

Exclusion Criteria:

* Neurologic and/or psychiatric known related disorders
* Malformation of the inner ear: the MRI scanners are routine examinations, in case of a cochlear implantation evaluation.
* Progressive or acquired deafness

Ages: 8 Months to 38 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2012-01; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Measurement of the score of perception of words in open list | 12 months after the implantation
  Measurement of the score of perception of words in open list in the noise 12 and 24 months after the implantation

SECONDARY OUTCOMES:
Measurement of the capability of localization right/left | 12 and 24 months after the implantation
  Measurement of the capability of localization right/left
Measurement of the level of comprehension and production | 24 months after the implantation
  Measurement of the level of comprehension and production after 24 months after the implantation
Evaluation of the medical monitoring about the materiovigilance and the eventual complications | During all the duration of the study
  Evaluation of the medical monitoring about the materiovigilance and the eventual complications
Measurement of the vestibulometry and of the children's psychomotor development | 12 and 24 months after the implantation
  Measurement of the vestibulometry and of the children's psychomotor development
Analysis of the parent questionnaires of the quality of life | 12 and 24 months after implantation
  Analysis of the parent questionnaires of the quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie Loundon, MD, MD-PhD, Principal Investigator — Assistance Publique